CLINICAL TRIAL: NCT06301854
Title: A Multicenter, Open Study to Evaluate the Long-term Safety and Efficacy of TPN171H in Patients With Erectile Dysfunction
Brief Title: Long-term Safety of TPN171H Tablet in Erectile Dysfunction.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPN171H-E302
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TPN171H group (Experimental): 10 mg/ time, as needed, it is recommended to take warm water within 0.5 to 4 hours before sexual activity.
  Interventions: Drug: TPN171H

INTERVENTIONS:
Drug: TPN171H — 10 mg/ time, as needed, it is recommended to take warm water within 0.5 to 4 hours before sexual activity.
  Other Names: Simmerafil

SUMMARY:
This is a multicenter, open study to evaluate the long-term safety and efficacy of TPN171H in men with erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 75 years (inclusive);
* Males with ED at least 3 months;
* IIEF-5 ≤ 21 at visit 1;
* Patients in a stable, heterosexual relationship during the study;
* At the end of the untreated baseline period, the following conditions are met：（1）The subject must make at least four attempts at sexual intercourse during the untreated baseline period. （2）At least 50% of attempts during this period must be unsuccessful,（unsuccess means at least one of the first three questions should be answered "No" in SEP）.（3）5≤IIEF-EF≤25.
* Patients who are willing to have 4 or more attempts of sexual intercourse per month, demonstrated compliance with the study protocol, including drug administration, diary completion, and scheduled study visits, during the qualifying trial;
* Patients who are willing to take proper contraceptive during the study and within 3 months after the last dose;
* Patients who have voluntarily decided to participate in this study, and signed the informed consent form.

Exclusion Criteria:

* Patients who have a history of hypersensitivity to other PDE5 inhibitors or TPN171H;
* Patients with anatomical malformations of the penis;
* Patients with primary hypoactive sexual desire;
* Patients with ED, which is caused by any other primary sexual disorder;
* Patients with ED, which is caused by spinal injury or have had a radical prostatectomy or other surgery;
* Patients who have a penile implant;
* Patients who do not respond to marketed PDE5 inhibitors or have adverse reactions that lead to drug discontinuation;
* CYP3A4 potent inhibitors, moderate inhibitors, and potent inducers need to be used during the trial or discontinued for less than 31 days before enrollment;
* Subjects who are taking nitrate or NO donor drugs, guanylate cyclase agonists and cannot be discontinued during the trial;
* Patients with the following cardiovascular disease: Myocardial infarction or stroke within the last 6 months; Unstable angina or angina occurring during sexual intercourse; New York Heart Association Class 2 or greater heart failure in the last 6 months;
* Uncontrolled hypotension (<90/60mmHg) or uncontrolled hypertension (≥180/110mmHg);
* Patients with diabetic complications (diabetic nephropathy, peripheral neuropathy);
* Patients with hepatic or renal dysfunction as per the following: AST, ALT>3*ULN, serum creatinine exceeds 50% of the upper limit of normal value;
* Patients with active gastrointestinal ulcers and bleeding disorders;
* Patients who have a history of NAION, or with a known genetically degenerative retinopathy, including retinitis pigmentosa;
* Patients who have a history of sudden decrease or loss of hearing;
* Patients with a history of severe central nervous system injury or peripheral muscular neurological disease in the past 6 months;
* Patient with a history of malignancy;
* Patients with significant neurological abnormalities who are unable or unwilling to cooperate;
* Patients whose partner is breastfeeding/pregnant/trying to become pregnant, has a gynecological disease or is restricted in their activities during treatment;
* Patients who have used other drugs in clinical trials within the last 1 month;
* For other reasons besides the aforementioned cases, patient whose participation is deemed inappropriate.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) and adverse drug reactions (ADRs) during treatment observation. | during the treatment and observation.
  Adverse events occurring throughout the study period were assessed and graded.

SECONDARY OUTCOMES:
Change From Baseline in the International Index of Erectile Function - Erectile Function. | baseline，3 months, 6 months
  The primary efficacy variable was the change in the EF domain scores of the IIEF questionnaire from baseline, calculated by comparing total scores from questions 1-5 and 15 from the IIEF questionnaire .
Change From Baseline in Question 2 of the Patient Sexual Encounter Profile (SEP) Diary at the 3rd and 6th month in Percentage of Yes Responses. | baseline，3 months, 6 months
  Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 2. "Were you able to insert your penis into your partner's vagina when you are trying to have sex ?" Data are presented as the mean percentage of yes responses per participant.
Change From Baseline in Question 3 of the Patient Sexual Encounter Profile (SEP) Diary at the 3rd and 6th month in Percentage of Yes Responsesat Week 12 in Percentage of Yes Responses. | baseline，3 months, 6 months
  Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 3. "Did your erection last long enough for you to have successful intercourse?" Data are presented as the mean percentage of yes responses per participant.
Percentage of subjects whose IIEF-EF scores returned to normal (≥26) at the 3rd and 6th month of medication. | baseline，3 months, 6 months
  Assessed was the changes in the number of subjects whose IIEF domain score at the 6th month visit was ≥26.
Change From Baseline to the 3rd months and 6th months Endpoint in International Index of Erectile Function (IIEF),Orgasmic Functions,Sexual Desire,Intercourse Satisfaction, Overall Satisfaction. | baseline，3 months, 6 months
  Self-reported, Orgasmic Functions, Sexual Desire, Intercourse Satisfaction, Overall Satisfaction.
Percentage of respondents who answered "yes" to questions 1 and 2 of the Comprehensive Evaluation Questionnaire (GAQ) at 3 Erectile Function (IIEF),Orgasmicand at the 3rd and 6th month. | 3 months, 6 months
  Percentage of respondents who answered "yes" to questions 1 and 2 of the GAQ. GAQ1: Has the treatment you have been taking during this study improved your erections? GAQ2: If yes, has the treatment improved your ability to engage in sexual activity? The data is expressed as the average percentage of "yes" answers per participant.
Change From Baseline in the International Index of Erectile Function - Erectile Function. | baseline，3 months, 6 months, 9 months and 12 months
  The primary efficacy variable was the change in the EF domain scores of the IIEF questionnaire from baseline, calculated by comparing total scores from questions 1-5 and 15 from the IIEF questionnaire .
Change From Baseline in Question 2 of the Patient Sexual Encounter Profile (SEP) Diary at the 3rd，6th，9th，12th month in Percentage of Yes Responses. | baseline，3 months, 6 months, 9 months and 12 months
  Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 2. "Were you able to insert your penis into your partner's vagina when you are trying to have sex ?" Data are presented as the mean percentage of yes responses per participant.
Change From Baseline in Question 3 of the Patient Sexual Encounter Profile (SEP) Diary at the 3rd，6th，9th，12th month in Percentage of Yes Responsesat Week 12 in Percentage of Yes Responses. | baseline，3 months, 6 months, 9 months and 12 months
  Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 3. "Did your erection last long enough for you to have successful intercourse?" Data are presented as the mean percentage of yes responses per participant.
Percentage of subjects whose IIEF-EF scores returned to normal (≥26) at the the 3rd，6th，9th，12th month of medication. | baseline，3 months, 6 months, 9 months and 12 months
  Assessed was the changes in the number of subjects whose IIEF domain score at the 3rd，6th，9th，12th month visit was ≥26.
Change From Baseline to the 3rd，6th，9th，12th month Endpoint in International Index of Erectile Function (IIEF),Orgasmic Functions,Sexual Desire,Intercourse Satisfaction, Overall Satisfaction. | baseline, 3 months, 6 months, 9 months and 12 months
  Self-reported, Orgasmic Functions, Sexual Desire, Intercourse Satisfaction, Overall Satisfaction.
Percentage of respondents who answered "yes" to questions 1 and 2 of the Comprehensive Evaluation Questionnaire (GAQ) at 3 Erectile Function (IIEF),Orgasmicand at the 3rd，6th，9th，12th month . | 3 months, 6 months, 9 months and 12 months
  Percentage of respondents who answered "yes" to questions 1 and 2 of the GAQ. GAQ1: Has the treatment you have been taking during this study improved your erections? GAQ2: If yes, has the treatment improved your ability to engage in sexual activity? The data is expressed as the average percentage of "yes" answers per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Jiang, Principal Investigator — Peking University First Hospital
Locations (34):
- China (34):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong
  - The Second Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Shenzhen Songgang People's Hospital, Shenzhen, Guangdong
  - The 2nd Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Qingyuan People's Hospital, Qingyuan, G
  - The Second Hospital of Hebei Medical Uniyersity, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University, Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Wuhan Union Hospital, Wuhan, Hubei
  - The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine, Changsha, Hunan
  - Loudi Central Hospital, Loudi, Hunan
  - Yueyang People's Hospital, Yueyang, Hunan
  - Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Nanchang reproductive hospital, Nanchang, Jiangxi
  - Yichang Central People's Hospital (Xiling Campus), Yichang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Chifeng Municipal Hospital, Chifeng, Neimenggu
  - The Affiliated Hospital of Qinghai University, Xining, Qinghai
  - Xianyang Central Hospital, Xianyang, Shanxi
  - The Second Affiliated Hospital of Shaanxi University of Chinese Medicine, Xian, Shanxi
  - Nuclear Industry 416 Hospital, Chengdu, Sichuang
  - The Affiliated Hospital of Chengdu University, Chengdu, Sichuang
  - Suining Central Hospital, Suining, Sichuang
  - Xinjiang Uygur Autonomous Region Hospital of Traditional Chinese Medicine, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No